CLINICAL TRIAL: NCT00003006
Title: Detection of Occult Micrometastases in Patients With Clinical Stage I NSCLC: A Prospective Analysis
Brief Title: Detection of Early Metastases in Patients With Stage I Non-small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-9761; U10CA031946 (NIH); CLB-9761; CDR0000065576 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2003-08-13 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Reverse Transcriptase Polymerase Chain Reaction; Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients enrolled onto CALGB 9761 will have, at the time of thoracotomy (or video assisted lobectomy) and pulmonary resection, samples of bone marrow, primary tumor, and intrathoracic lymph nodes harvested.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: At the time of thoracotomy and pulmonary resection, patients have samples of bone marrow, primary tumor, and intrathoracic lymph nodes harvested. The presence of occult metastases in bone marrow and lymph nodes is assessed using immunohistochemistry or reverse transcriptase-polymerase chain reaction.
  Interventions: Genetic: reverse transcriptase-polymerase chain reaction; Other: immunohistochemistry staining method

INTERVENTIONS:
Genetic: reverse transcriptase-polymerase chain reaction
Other: immunohistochemistry staining method

SUMMARY:
RATIONALE: Detecting very early metastases in bone marrow and/or lymph nodes may help doctors plan better treatment for non-small cell lung cancer.

PURPOSE: Clinical trial to detect the presence of metastatic cancer in patients with stage I non-small cell lung cancer that has not been previously treated.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether the presence of occult micrometastases (OM) detected by immunohistochemistry or reverse transcriptase-polymerase chain reaction (RT-PCR) in histologically negative lymph nodes or bone marrow is associated with poorer survival among patients with stage I non-small cell lung cancer.
* Determine the incidence of OM in histologically negative lymph nodes and bone marrow by immunohistochemistry (staining for cytokeratins and the CEA glycoprotein) or RT-PCR (to detect CEA mRNA) in these patients.
* Assess the sensitivity of immunohistochemistry relative to RT-PCR for detecting OM in these patients.
* Determine the relationship between tumor size (or T-stage) and the presence of OM detected by immunohistochemistry or RT-PCR in these patients.
* Determine the relationship between the presence of OM and disease-free survival in these patients.
* Determine the relationship between the site of OM and incidence of recurrence, site of recurrence, and survival of these patients.

OUTLINE: At the time of thoracotomy and pulmonary resection, patients have samples of bone marrow, primary tumor, and intrathoracic lymph nodes harvested. The presence of occult metastases in bone marrow and lymph nodes is assessed using immunohistochemistry or reverse transcriptase-polymerase chain reaction.

Patients are followed every 6 months for 5 years.

ELIGIBILITY:
* Clinical stage I proven or suspected new non-small cell lung carcinoma T1 or T2 primary N1 or N2 lymph nodes <1cm on CT or negative mediastinoscopy
* ≥ 5 years since prior chemo or XRT; no prior mediastinal or chest XRT.
* ≥ 18 years of age
* No history of previous lung cancer or concomitant malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-small cell lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 1997-05; Primary Completion 2002-03 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
overall survival | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Maddaus, MD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (10):
- United States (10):
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina

REFERENCES:
- [Background] Potti A, Mukherjee S, Petersen R, Dressman HK, Bild A, Koontz J, Kratzke R, Watson MA, Kelley M, Ginsburg GS, West M, Harpole DH Jr, Nevins JR. A genomic strategy to refine prognosis in early-stage non-small-cell lung cancer. N Engl J Med. 2006 Aug 10;355(6):570-80. doi: 10.1056/NEJMoa060467. PMID 16899777 (Retraction: PMID 21366430 Potti A, Mukherjee S, Petersen R, Dressman HK, Bild A, Koontz J, Kratzke R, Watson MA, Kelley M, Ginsburg GS, West M, Harpole DH Jr, Nevins JR. N Engl J Med. 2011 Mar 24;364(12):1176)
- [Result] Maddaus MA, Wang X, Vollmer RT, et al.: CALGB 9761: a prospective analysis of IHC and PCR based detection of occult metastatic disease in stage I NSCLC. [Abstract] J Clin Oncol 24 (Suppl 18): A-7030, 371s, 2006.
- [Result] D'Cunha J, Herndon JE 2nd, Herzan DL, Patterson GA, Kohman LJ, Harpole DH, Kernstine KH, Kern JA, Green MR, Maddaus MA, Kratzke RA; Cancer and Leukemia Group B. Poor correspondence between clinical and pathologic staging in stage 1 non-small cell lung cancer: results from CALGB 9761, a prospective trial. Lung Cancer. 2005 May;48(2):241-6. doi: 10.1016/j.lungcan.2004.11.006. Epub 2005 Jan 4. PMID 15829324
- [Result] D'Cunha J, Herndon JL, Herzan DL, et al.: Poor correlation between clinical and pathological staging in stage I non-small cell lung cancer: results from CALGB 9761, a prospective trial. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-2550, 634, 2003.
- [Result] Vollmer RT, Herndon JE 2nd, D'Cunha J, Abraham NZ, Solberg J, Fatourechi M, Maruska A, Kern JA, Green MR, Kratzke RA, Maddaus MA; Cancer and Leukemia Group B Trial 9761. Immunohistochemical detection of occult lymph node metastases in non-small cell lung cancer: anatomical pathology results from Cancer and Leukemia Group B Trial 9761. Clin Cancer Res. 2003 Nov 15;9(15):5630-5. PMID 14654545
- [Result] D'Cunha J, Corfits AL, Herndon JE 2nd, Kern JA, Kohman LJ, Patterson GA, Kratzke RA, Maddaus MA. Molecular staging of lung cancer: real-time polymerase chain reaction estimation of lymph node micrometastatic tumor cell burden in stage I non-small cell lung cancer--preliminary results of Cancer and Leukemia Group B Trial 9761. J Thorac Cardiovasc Surg. 2002 Mar;123(3):484-91; discussion 491. doi: 10.1067/mtc.2002.119883. PMID 11882819